CLINICAL TRIAL: NCT00813930
Title: Lifestyle Intervention For Effective Diabetes Management (LIFE-DM) Trial
Brief Title: Lifestyle Intervention For Effective Diabetes Management
Acronym: LIFE-DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: St. Joseph's Health Centre Toronto (Other); University Health Network, Toronto (Other)
Responsible Party: Dr. Gillian Booth, St. Michael's Hospital, Toronto
Allocation: Randomized | Model: Parallel | Purpose: Supportive Care
Other Study IDs: SMH-LKSKI
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2010-03-23 (Estimated); Status verified 2010-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Lifestyle Intervention; Cardiovascular risk reduction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- INTERxVENT Program (Experimental): Participants in INTERxVENT will complete a 'Baseline Assessment' and 'Follow-up' questionnaire, and will have a health professional visit his/her home for an initial assessment (BP,height,weight,waist measurement) and blood collection (blood glucose and cholesterol levels). As part of the program, each participant will also complete a self-reported 'Health History Questionnaire' (HHQ); a follow-up HHQ will be completed about 12 weeks into the program to monitor progress. Each participant randomized to INTERxVENT receives educational articles which address diabetes management issues. A structured, individualized program, consisting of educational materials and 12 live mentoring/coaching telephone calls will take place over 6 months. The mentors consist of allied health professionals. The sequence by which educational content is administered will be both self-directed and guided by the mentors using an algorithmic approach according to the participant's readiness-to-change scores.
  Interventions: Behavioral: INTERxVENT lifestyle modification program
- Usual medical care (No Intervention): Each participant randomized to this group will not receive any formal intervention but will receive the same care over the 6-month period as he/she usually receives from his/her health care team. Participants in this group will undergo the same baseline and outcome assessment as those in the intervention group, including blood pressure (BP) measurement, physical assessment (height, weight, waist measurement) and blood collection (blood glucose and cholesterol levels), as well as completion of the 'Baseline Assessment' and 'Follow-up' questionnaires.

INTERVENTIONS:
Behavioral: INTERxVENT lifestyle modification program — It is a lifestyle behavior modification program which helps Type 2 diabetics manage diabetes better and reduce cardiovascular risk factors. The program involves up to 12 telephone mentor/coaching sessions with a certified health professional.
  Other Names: INTERxVENT
  Arms: INTERxVENT Program

SUMMARY:
Chronic disease management programs are shown to reduce mortality, recurrent hospitalizations, and improve indirect societal costs among specific subgroups of the population. INTERxVENT is one such individualized chronic cardiovascular and lifestyle management program, comprised of several individualized modules - diet, exercise, stress management, smoking cessation, chronic disease - prescribed algorithmically according to patient risk profile, environmental surroundings, and behavioural readiness-to-change. Nonrandomized studies assessing INTERxVENT in diabetic, pre-diabetic, and metabolic syndrome populations have demonstrated improvement in several intermediary endpoints, including reductions in fasting glucose, lipids, and blood pressure. However, no randomized controlled clinical trials in these populations have been conducted. This pilot study is a randomized clinical trial evaluating the effectiveness of INTERxVENT as compared with 'usual medical care' in improving cardiovascular risk-factor profiles among individuals with diabetes. Additionally, the extent to which such findings are generalizable to diabetic, socially vulnerable, populations is unknown, thus this will be examined also.

DETAILED DESCRIPTION:
Diabetes is a leading cause of cardiovascular mortality and morbidity, and is more often than not a very difficult disease for individuals to manage effectively. People with diabetes have to be committed to a self-care regimen which includes, careful monitoring of blood sugar, blood pressure, cholesterol, eating healthy, exercising, foot care and regular physical and eye check-ups. This can be quite daunting and stressful for some to undertake themselves, and is largely dependent on individual self-motivation. Family physicians assist their patients in managing their diabetes but they have significant time constraints and may not always be able to deliver the high service intensity required to reduce morbidity and/or may have inadequate access to resources to help patients positively change their self-care behaviour.

Chronic disease-management programs involving home-based nursing health promotion have been shown to reduce mortality, reduce recurrent hospitalization, and improve indirect societal costs among specific subgroups of the population, including those with diabetes, however, such interventions can be costly and cumbersome to implement given the need for home-based visits.

INTERxVENT is a telephone-based, individualized, chronic cardiovascular and lifestyle management program combining a formal management plan, case-managed care (through a coach/mentor), and educational modules to teach patients to modify and sustain healthy lifestyle behaviours. It is comprised of several individualized modules (e.g., diet, exercise, stress management, smoking cessation, chronic disease), which are prescribed algorithmically in accordance to a patient's individual risk profile, environmental surroundings, and behavioural readiness to change. All recommendations are according to best-practice standards and evidence-based guidelines.

Nonrandomized intervention studies assessing INTERxVENT in diabetic, pre-diabetic, and metabolic syndrome populations have demonstrated significant reductions in biologically relevant measures, such as fasting glucose, glycosylated hemoglobin (HbA1c), lipids, and blood pressure. However, no randomized controlled clinical trials in these populations assessing the impact of INTERxVENT have been conducted.

The proposed pilot study will evaluate the efficacy of INTERxVENT as compared with 'usual medical care' in improving cardiovascular risk-factor profiles among individuals with diabetes. In addition, to what extent a chronic disease management program will yield similar effectiveness in socio-economically disadvantaged individuals is unknown. We hypothesize that chronic disease management programs, like INTERxVENT, will result in improved intermediary biological and behavioural risk profiles for all program participants randomized to this intervention, regardless of socio-economic condition.

The results of this pilot study will determine and assist in designing and ascertaining sample sizes for a larger trial, respectively, should such a trial be warranted. Additionally, such chronic disease management interventions may improve the overall health of partaking individuals and relieve strain and decrease costs within the existing health care system.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Age 18 years or older

Exclusion Criteria:

* Documented history of myocardial infarction, stroke, angina, angioplasty, or bypass surgery
* Unable to understand written and spoken English
* Presence of cognitive impairment (e.g., dementia) or significant psychological problems (e.g., schizophrenia, schizoaffective disorders) that, in the investigators' opinion, may prohibit the participant from following study protocols
* Unavailable to participate (e.g., incarceration, no access to a telephone)
* HIV / AIDS
* Estimated life expectancy less than one year in the opinion of the clinician
* Participation in any other clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Six-month United Kingdom Prospective Diabetes Study (UKPDS) risk engine score. The UKPDS risk engine is a validated scoring system that uses multiple clinical characteristics to predict new coronary heart disease risks in patients with type 2 diabetes. | 6 months

SECONDARY OUTCOMES:
Six-month: HbA1c, seated systolic blood pressure, serum Total Cholesterol concentration, serum HDL-C concentration, Total/HDL-C ratio value, LDL-C concentration, self-reported smoking status, adherence to medications and lifestyle measures. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gillian L. Booth, MD, MSc, Principal Investigator — Li Ka Shing Knowledge Institute, St. Michael's Hospital
Locations (3):
- Canada (3):
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto Western Hospital, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario

REFERENCES:
- [Background] Booth GL, Kapral MK, Fung K, Tu JV. Recent trends in cardiovascular complications among men and women with and without diabetes. Diabetes Care. 2006 Jan;29(1):32-7. doi: 10.2337/diacare.29.01.06.dc05-0776. PMID 16373892
- [Background] Booth GL, Kapral MK, Fung K, Tu JV. Relation between age and cardiovascular disease in men and women with diabetes compared with non-diabetic people: a population-based retrospective cohort study. Lancet. 2006 Jul 1;368(9529):29-36. doi: 10.1016/S0140-6736(06)68967-8. PMID 16815377
- [Background] Simpson SH, Corabian P, Jacobs P, Johnson JA. The cost of major comorbidity in people with diabetes mellitus. CMAJ. 2003 Jun 24;168(13):1661-7. PMID 12821619
- [Background] Bonow RO, Gheorghiade M. The diabetes epidemic: a national and global crisis. Am J Med. 2004 Mar 8;116 Suppl 5A:2S-10S. doi: 10.1016/j.amjmed.2003.10.014. PMID 15019858
- [Background] Buhrmann R, Asaad D, Hux JE, Tang M, Sykora K: Diabetes and the Eye. In Diabetes in Ontario: an ICES practice atlas. Hux JE, Booth GL, Slaughter P, Laupacis A, Eds. Toronto, Institute for Clinical Evaluative Sciences, 2003.
- [Background] Shah BR, Mamdani M, Kopp A: Drug Use in Older People with Diabetes. In Diabetes in Ontario: an ICES practice atlas. Hux JE, Booth GL, Slaughter P, Laupacis A, Eds. Toronto, Insitute for Clinical Evaluative Sciences, 2003.
- [Background] Markle-Reid M, Weir R, Browne G, Roberts J, Gafni A, Henderson S. Health promotion for frail older home care clients. J Adv Nurs. 2006 May;54(3):381-95. doi: 10.1111/j.1365-2648.2006.03817.x. PMID 16629922
- [Background] Markle-Reid M, Browne G, Weir R, Gafni A, Roberts J, Henderson SR. The effectiveness and efficiency of home-based nursing health promotion for older people: a review of the literature. Med Care Res Rev. 2006 Oct;63(5):531-69. doi: 10.1177/1077558706290941. PMID 16954307
- [Background] Gordon NF, Salmon RD, Mitchell BS, Faircloth GC, Levinrad LI, Salmon S, Saxon WE, Reid KS. Innovative approaches to comprehensive cardiovascular disease risk reduction in clinical and community-based settings. Curr Atheroscler Rep. 2001 Nov;3(6):498-506. doi: 10.1007/s11883-001-0040-9. PMID 11602070
- [Background] Gordon NF, English CD, Contractor AS, Salmon RD, Leighton RF, Franklin BA, Haskell WL. Effectiveness of three models for comprehensive cardiovascular disease risk reduction. Am J Cardiol. 2002 Jun 1;89(11):1263-8. doi: 10.1016/s0002-9149(02)02323-8. PMID 12031725
- [Background] Gordon NF, Salmon RD, Franklin BA, Sperling LS, Hall L, Leighton RF, Haskell WL. Effectiveness of therapeutic lifestyle changes in patients with hypertension, hyperlipidemia, and/or hyperglycemia. Am J Cardiol. 2004 Dec 15;94(12):1558-61. doi: 10.1016/j.amjcard.2004.08.039. PMID 15589017
- [Background] Stevens RJ, Kothari V, Adler AI, Stratton IM; United Kingdom Prospective Diabetes Study (UKPDS) Group. The UKPDS risk engine: a model for the risk of coronary heart disease in Type II diabetes (UKPDS 56). Clin Sci (Lond). 2001 Dec;101(6):671-9. PMID 11724655